CLINICAL TRIAL: NCT00674778
Title: Prospective Registry on Vascular Access in Interventions in Lazio Region
Acronym: PREVAIL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: San Filippo Neri General Hospital (Other)
Responsible Party: Christian Pristipino, MD, San Filippo Neri Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1/6/2006
Record Dates: First submitted 2008-05-05; First posted 2008-05-08 (Estimated); Last update posted 2008-05-08 (Estimated); Status verified 2008-05

CONDITIONS: Postoperative Hemorrhages
Keywords: Radial; Femoral; artery; Invasive cardiology safety
MeSH Terms: conditions — Postoperative Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Radial approach
  Interventions: Procedure: Any percutaneous cardiovascular procedure
- 2 (Active Comparator): Femoral approach
  Interventions: Procedure: Any percutaneous cardiovascular procedure

INTERVENTIONS:
Procedure: Any percutaneous cardiovascular procedure

SUMMARY:
Previous randomised studies showed that radial artery catheterisation for percutaneous cardiovascular procedures has a superior safety profile than femoral access, however the confirmation of these benefits in the real world by a large, specific, observational study is still lacking.

We endeavoured to assess the access site-related outcomes of any percutaneous cardiovascular procedure by designing a prospective registry monitoring a consecutive sample of patients in a short period of time at nine Roman hospitals reflecting the contemporary state of health care.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing any percutaneous cardiovascular procedure

Exclusion Criteria:

* Patients already enrolled in other clinical trials

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1052 (Actual)
Dates: Start 2006-06; Study Completion 2006-06

PRIMARY OUTCOMES:
Cumulative incidence of: (a) major and minor bleedings, (b) access site vascular complications, (c) stroke | in-hospital

SECONDARY OUTCOMES:
Cumulative incidence of (a) death, (b) myocardial infarction or reinfarction | in-hospital

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Richichi, MD, Study Chair — San Filippo Neri Hospital